CLINICAL TRIAL: NCT06542770
Title: Subtle Ultrasound Atrial Anomalies Predicts the Early Diagnosis of Silent Atrial Fibrillation Detected by Implantable Cardiac Monitor in Patients With Cryptogenic Stroke. A Randomized Trial
Brief Title: Atrial Anomalies Predict Silent Atrial Fibrillation Detected by Implantable Cardiac Monitor in Cryptogenic Stroke
Acronym: CRIPTO-FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Ermengol Vallès, Head of arrhythmias, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRIPTO-FAST
Record Dates: First submitted 2024-07-21; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Atrial Fibrillation; Cardiac Rhythm Disorder; Left Atrial Dilatation; Cryptogenic Stroke
Keywords: Atrial strain. Implantable cardiac monitor
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Randomized prospective parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Atrial cardiomyopathy by echocardiogram intervention (Experimental): Presence of Atrial cardiomyopathy is defined by echocardiogram if ANY of the following is present:
  1. LA dilatation: indexed volumen >32 ml/m2
  2. PALS (Peak atrial longitudinal strain) <21%
  3. PACS ( Peak atrial contraction strain ) <13%
  4. Atrial ejection fraction <55%
  Interventions: Device: Early implant of cardiac monitor
- Atrial cardiomyopathy by echocardiogram standard practice (No Intervention): Presence of Atrial cardiomyopathy is defined by echocardiogram if ANY of the following is present:
  1. LA dilatation: indexed volumen >32 ml/m2
  2. PALS (Peak atrial longitudinal strain) <21%
  3. PACS ( Peak atrial contraction strain ) <13%
  4. Atrial ejection fraction <55%
- Non atrial cardiomyopathy by echocardiogram intervention (Experimental): Absence of atrial cardiomyopathy is defined by echocardiogram if none of the characteristics bellow were accomplished.
  1. LA dilatation: indexed volumen >32 ml/m2
  2. PALS (Peak atrial longitudinal strain) <21%
  3. PACS ( Peak atrial contraction strain ) <13%
  4. Atrial ejection fraction <55%
  Interventions: Device: Early implant of cardiac monitor
- Non atrial cardiomyopathy by echocardiogram standard practice (No Intervention): Absence of atrial cardiomyopathy defined by echocardiogram if none of the characteristics bellow were accomplished.
  1. LA dilatation: indexed volumen >32 ml/m2
  2. PALS (Peak atrial longitudinal strain) <21%
  3. PACS ( Peak atrial contraction strain ) <13%
  4. Atrial ejection fraction <55%

INTERVENTIONS:
Device: Early implant of cardiac monitor — ICM implant 3-4 days after the stroke and prior to discharge. All devices (Abbott Confirm or Jot) were implanted subcutaneously under local anaesthesia in the left chest region and programmed with an specific algorithm for AF detection set at 30 seconds for detection. All patients were included in remote monitoring system (Merlin), which was programmed to send alerts in case of registering episodes qualifying for AF detection, and a monthly routine registration. All ICM recordings were reviewed by a specialized cardiologist.
  Arms: Atrial cardiomyopathy by echocardiogram intervention; Non atrial cardiomyopathy by echocardiogram intervention

SUMMARY:
Cryptogenic stroke (CS) causes about 30% of admissions to a stroke unit. Silent paroxysmal atrial fibrillation (PAF) is believed to be the underlying cause of a significant proportion of patients. The use of implantable cardiac monitors (ICM) early after the CS has demonstrated benefits in the diagnostic yield, but the indication for ICM in the current guidelines remains unclear. Atrial contraction strain (ACS) evaluated by cardiac ultrasound could be of help to select the patients more prone to suffer from silent PAF.

The purpose of this investigation is to conduct a randomized prospective unicentric study to evaluate the usefulness of ICM for early detection of silent PAF episodes in patients with CS. Clinical and ultrasound predictors of PAF occurrence (ACS) will be studied in order to define patients needing a closer follow-up.

DETAILED DESCRIPTION:
Introduction

Cryptogenic stroke (CS) is a stroke in which etiology cannot be determined after a comprehensive evaluation and it is the cause of about 30% of admissions to a stroke unit. In these cases single antiplatelet therapy is recommended as a long term treatment. However, silent paroxysmal atrial fibrillation (PAF) is believed to be the underlying cause of a significant proportion of episodes, and it´s recognition merits urgency since carries to oral anticoagulation (OAC) and antiplatelet therapy cessation. According to guidelines, in order to detect PAF we need to monitor the patient´s ECG for at least 48h, although the longer the monitoring is, the better the diagnostic yield.

Previous research showed controversial results regarding the use of implantable cardiac monitors (ICM) in such patients when the ICM had been implanted late after the CS. On the other hand, studies with an early implant demonstrated a clear benefit in the diagnostic yield. To date, the strategy to search actively for PAF in patients with CS is still not well established, and even when internal loop recorders (ILR) are our best option to recognize paroxysmal arrhythmic events, guidelines are not clear about the cases in which they might be indicated. Some markers, such as age, cardiovascular risk factors, blood biomarkers or cardiac ultrasound characteristics have been related to a higher silent PAF detection. Recent data points at the use of left atrium atrial strain (LAS) to select the patients more prone to suffer from silent PAF.

It remains to be defined the usefulness of ILR implanted early after the CS in order to diagnose the presence of silent PAF, and the roll or ACS in such patients in order to predict those being at higher risk.

Methods

This is a randomized prospective unicentric study to evaluate the usefulness of ICM for early detection of silent PAF episodes in patients with CS. During the first 48 hours from admission, patients were randomized to receive standard care (Control Group) or early ICM implantation (Study Group) before discharge. A special effort will be made to search for the clinical and ultrasound atrial predictors of PAF occurrence in order to better define what patients need a closer follow-up.

Ultrasound evaluation

The following ultrasound atrial features will be studied to separate patients into two categories:

1. LA dilatation: indexed volumen >32 ml/m2
2. PALS (Peak atrial longitudinal strain) <21%
3. PACS ( Peak atrial contraction strain ) <13%
4. Atrial ejection fraction <55%

Patients will be considered as having a "normal" LA if none of the above mentioned characteristics is accomplished, in opposition to patients who accomplish at least one characteristic described above, which will be considered as "atrial cardiomyopathy" patients.

Patients will be immediately treated with antiplatelet treatment. OAC will be started if PAF is detected during admission. Whilst in the Stroke Unit, all patients will be continuously ECG-monitored for at least 48 h and will undergo a cardiac transthoracic echocardiogram with complete evaluation of strain parameters.

Demographic factors, vascular risk factors and comorbidities will be collected. Work-up during admission will include, at least, a complete neurological examination, 12-lead ECG, brain computed tomography (CT), blood test and neurovascular imaging (magnetic resonance angiography, angioCT and/or two-dimensional ultrasound of supra-aortic trunks and intracranial territory).

The diagnosis of CS will be revisited in all patients 3 months after the index episode, and those found to have any potential cause other than PAF will be additionally excluded. The study follows national and international principles (Declaration of Helsinki), and it was approved by the local ethics committee. All patients are required to sign the specific informed consent.

Strategies for PAF detection Since the prevalence of AF is higher in patients having LA anomalies, we will divide the total group into two categories before randomization, depending on the presence or absence of: LA dilatation, and/or impaired ACS. Then we will randomize all patients to Control Group or Study Group.

Control group: after discharge from the Stroke Unit, patients in the control group will be studied with daily ECGs whilst admitted at the hospital. Outpatient serial ECGs will be performed at the time of each visit at the Neurology Clinic 3, 6 and 12 months after the stroke, and every 6 months thereafter. Additional ECGs will be performed if patients had symptoms potentially related to PAF. Furthermore all patients will undergo a 72h-Holter-monitoring scheduled 1 month after discharge.

Study group: patients in the active study group will undergo an ICM implant 3-4 days after the stroke and prior to discharge. All devices (Abbott Jot) will be implanted subcutaneously under local anaesthesia in the left chest region and programmed with an specific algorithm for AF detection set at 30 seconds for detection. All patients will be included in remote monitoring system (Merlin), which will be programmed to send alerts in case of registering episodes qualifying for AF detection, and a monthly routine registration. All ICM recordings will be reviewed by a specialized cardiologist. Patients will be seen at the arrhythmia and the neurology outpatient clinics at 3, 6 and 12 months after the stroke, and every 6 months thereafter.

End-points and follow-up Primary clinical outcome: detection of AF at follow-up, which is defined by the presence of a confirmatory 12-leads ECG, or a registration lasting more than 30 seconds in, either the 72h-Holter-Monitoring, or in the ICM recording. In case of AF detection OAC will be initiated immediately.

Secondary clinical outcomes: ultrasounds predictors for AF occurrence: LA indexed volumen, maximum systolic global longitudinal strain (PALs), atrial contraction strain (PACs), atrial ejection fraction.

We also will search for stroke recurrences, defined as new neurological events recorded after hospital discharge and validated by a vascular neurologist.

Statistical analysis Results are reported as mean (SD), median (p25-p75) or frequency (%). Comparisons between groups were performed with the Student t test or chi-squared analysis. The association between clinical variables and the study end-points was evaluated using survival analysis methodology (Cox regression models). The Kaplan-Meier method was used to estimate the cumulative probability of PAF detection and stroke recurrence in both groups, and comparisons were made by the log-rank test. Significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke or transient ischemic attack (TIA) from January 2022 to July 2023
* Age between 50 and 89 years;
* Undetermined origin at hospital admission according to the SSS-TOAST criteria (2):

  1. Absence of major structural heart disease by cardiac ultrasound (normal global and segmental left ventricle contraction, absence of valvular/rheumatic disease, absence of intracardiac shunts)
  2. Absence of AF during 48h ECG-monitoring
  3. Absence of major anomalies in the supra-aortic trunks ultrasound.

Exclusion Criteria:

1. Patients with a history of hemorrhagic stroke;
2. Presence with prior atrial fibrillation or atrial flutter;
3. Permanent contraindication or indication for OAC for other reasons;
4. Recent (<1 month) major surgery or cardiac events;
5. Presence of severe cardiac abnormalities;
6. Patients with life expectancy <1 year or severe stroke (modified Rankin Scale > 4).

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection atrial fibrilation at follow-up | Up to 2 years follow-up (ICM and standard care practice)
  defined by the presence of a confirmatory 12-leads ECG, or a registration lasting more than 30 seconds in, either the 72h-Holter-Monitoring, or in the ICM recording. In case of AF detection OAC was initiated immediately.

SECONDARY OUTCOMES:
LA indexed volume | Before Day 3 since the Criptogenic Stroke
  LA indexed volume in ml/m2
Maximum Systolic Global Longitudinal Strain (PALs) | Before Day 3 since the Criptogenic Stroke
  Maximum Systolic Global Longitudinal Strain (PALs) in %
Atrial Contraction Strain (PACs) | Before Day 3 since the Criptogenic Stroke
  atrial contraction strain (PACs) in %
Atrial Ejection Fraction | Before Day 3 since the Criptogenic Stroke
  Atrial ejection fraction in %
stroke recurrences | Up to 2 years follow-up (ICM and standard care practice)
  new neurological events recorded after hospital discharge and validated by a vascular neurologist

CONTACTS AND LOCATIONS:
Overall Officials: Ermengol Valles Gras, PhD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data from this study, including pseudoanonimized data from ultrasound exams and ECG signals from ICM will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the publication and during 10 years
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Andrew NE, Thrift AG, Cadilhac DA. The prevalence, impact and economic implications of atrial fibrillation in stroke: what progress has been made? Neuroepidemiology. 2013;40(4):227-39. doi: 10.1159/000343667. Epub 2013 Jan 24. PMID 23364221
- [Background] Sposato LA, Cipriano LE, Saposnik G, Ruiz Vargas E, Riccio PM, Hachinski V. Diagnosis of atrial fibrillation after stroke and transient ischaemic attack: a systematic review and meta-analysis. Lancet Neurol. 2015 Apr;14(4):377-87. doi: 10.1016/S1474-4422(15)70027-X. Epub 2015 Mar 4. PMID 25748102
- [Background] Rubiera M, Aires A, Antonenko K, Lemeret S, Nolte CH, Putaala J, Schnabel RB, Tuladhar AM, Werring DJ, Zeraatkar D, Paciaroni M. European Stroke Organisation (ESO) guideline on screening for subclinical atrial fibrillation after stroke or transient ischaemic attack of undetermined origin. Eur Stroke J. 2022 Sep;7(3):VI. doi: 10.1177/23969873221099478. Epub 2022 Jun 3. PMID 36082257
- [Background] Cuadrado-Godia E, Benito B, Ois A, Valles E, Rodriguez-Campello A, Giralt-Steinhauer E, Cabrera S, Alcalde O, Jimenez-Lopez J, Jimenez-Conde J, Marti-Almor J, Roquer J. Ultra-early continuous cardiac monitoring improves atrial fibrillation detection and prognosis of patients with cryptogenic stroke. Eur J Neurol. 2020 Feb;27(2):244-250. doi: 10.1111/ene.14061. Epub 2019 Sep 18. PMID 31424609
- [Background] Klijn CJ, Paciaroni M, Berge E, Korompoki E, Korv J, Lal A, Putaala J, Werring DJ. Antithrombotic treatment for secondary prevention of stroke and other thromboembolic events in patients with stroke or transient ischemic attack and non-valvular atrial fibrillation: A European Stroke Organisation guideline. Eur Stroke J. 2019 Sep;4(3):198-223. doi: 10.1177/2396987319841187. Epub 2019 Apr 9. PMID 31984228
- [Background] Pagola J, Juega J, Francisco-Pascual J, Bustamante A, Penalba A, Pala E, Rodriguez M, De Lera-Alfonso M, Arenillas JF, Cabezas JA, Moniche F, de Torres R, Montaner J, Gonzalez-Alujas T, Alvarez-Sabin J, Molina CA; Crypto-AF study group. Predicting Atrial Fibrillation with High Risk of Embolization with Atrial Strain and NT-proBNP. Transl Stroke Res. 2021 Oct;12(5):735-741. doi: 10.1007/s12975-020-00873-2. Epub 2020 Nov 13. PMID 33184686
- [Background] Albers GW, Bernstein RA, Brachmann J, Camm J, Easton JD, Fromm P, Goto S, Granger CB, Hohnloser SH, Hylek E, Jaffer AK, Krieger DW, Passman R, Pines JM, Reed SD, Rothwell PM, Kowey PR. Heart Rhythm Monitoring Strategies for Cryptogenic Stroke: 2015 Diagnostics and Monitoring Stroke Focus Group Report. J Am Heart Assoc. 2016 Mar 15;5(3):e002944. doi: 10.1161/JAHA.115.002944. No abstract available. PMID 27068633
- [Background] Rubio Campal JM, Garcia Torres MA, Sanchez Borque P, Navas Vinagre I, Zamarbide Capdepon I, Miracle Blanco A, Bravo Calero L, Saez Pinel R, Tunon Fernandez J, Serratosa Fernandez JM. Detecting Atrial Fibrillation in Patients With an Embolic Stroke of Undetermined Source (from the DAF-ESUS registry). Am J Cardiol. 2020 Feb 1;125(3):409-414. doi: 10.1016/j.amjcard.2019.10.050. Epub 2019 Nov 6. PMID 31780074
- [Background] Marks D, Ho R, Then R, Weinstock JL, Teklemariam E, Kakadia B, Collins J, Andriulli J, Hunter K, Ortman M, Russo AM. Real-world experience with implantable loop recorder monitoring to detect subclinical atrial fibrillation in patients with cryptogenic stroke: The value of p wave dispersion in predicting arrhythmia occurrence. Int J Cardiol. 2021 Mar 15;327:86-92. doi: 10.1016/j.ijcard.2020.11.019. Epub 2020 Nov 10. PMID 33186666
- [Background] Chorin E, Peterson C, Kogan E, Barbhaiya C, Aizer A, Holmes D, Bernstein S, Schole M, Duraiswami H, Spinelli M, Park D, Chinitz L, Jankelson L. Comparison of the Effect of Atrial Fibrillation Detection Algorithms in Patients With Cryptogenic Stroke Using Implantable Loop Recorders. Am J Cardiol. 2020 Aug 15;129:25-29. doi: 10.1016/j.amjcard.2020.05.027. Epub 2020 May 23. PMID 32600783
- [Background] Magnusson P, Lyren A, Mattsson G. Diagnostic yield of chest and thumb ECG after cryptogenic stroke, Transient ECG Assessment in Stroke Evaluation (TEASE): an observational trial. BMJ Open. 2020 Sep 24;10(9):e037573. doi: 10.1136/bmjopen-2020-037573. PMID 32973062
- [Background] Lumikari TJ, Putaala J, Kerola A, Sibolt G, Pirinen J, Pakarinen S, Lehto M, Nieminen T. Continuous 4-week ECG monitoring with adhesive electrodes reveals AF in patients with recent embolic stroke of undetermined source. Ann Noninvasive Electrocardiol. 2019 Sep;24(5):e12649. doi: 10.1111/anec.12649. Epub 2019 May 2. PMID 31045315
- [Background] Kalani R, Bernstein R, Passman R, Curran Y, Ruff I, Prabhakaran S. Factual Inaccuracies Contained in the Article Entitled "Low Yield of Mobile Cardiac Outpatient Telemetry after Cryptogenic Stroke in Patients with Extensive Cardiac Imaging". J Stroke Cerebrovasc Dis. 2017 Dec;26(12):3035. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.018. Epub 2017 Oct 18. No abstract available. PMID 29054732
- [Background] Ziegler PD, Rogers JD, Ferreira SW, Nichols AJ, Richards M, Koehler JL, Sarkar S. Long-term detection of atrial fibrillation with insertable cardiac monitors in a real-world cryptogenic stroke population. Int J Cardiol. 2017 Oct 1;244:175-179. doi: 10.1016/j.ijcard.2017.06.039. Epub 2017 Jun 10. PMID 28624331
- [Background] Ziegler PD, Rogers JD, Ferreira SW, Nichols AJ, Sarkar S, Koehler JL, Warman EN, Richards M. Real-World Experience with Insertable Cardiac Monitors to Find Atrial Fibrillation in Cryptogenic Stroke. Cerebrovasc Dis. 2015;40(3-4):175-81. doi: 10.1159/000439063. Epub 2015 Aug 28. PMID 26314298